CLINICAL TRIAL: NCT01114724
Title: Valiant® Thoracic Stent Graft With the Captivia Delivery System. Evaluation of the Clinical Performance of the Valiant Thoracic Stent Graft With the Captivia Delivery System (Valiant Captivia) for the Treatment of Acute, Complicated Type B Aortic Dissections
Brief Title: Study to Evaluate the Clinical Performance of the Valiant Thoracic Stent Graft With the Captivia Delivery System (Valiant Captivia) for the Treatment of Acute, Complicated Type B Aortic Dissections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP # 118
Record Dates: First submitted 2010-04-26; First posted 2010-05-03 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Aortic Dissection
Keywords: Thoracic dissection; Endovascular aortic repair
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valiant Thoracic Stent Graft with the Captivia Delivery System (Experimental)
  Interventions: Device: Valiant Thoracic Stent Graft with the Captivia Delivery System

INTERVENTIONS:
Device: Valiant Thoracic Stent Graft with the Captivia Delivery System — All subjects will be implanted with this device

SUMMARY:
The purpose of this study is to determine if the Valiant stent graft is safe and effective in treating patients who have a thoracic dissection. A thoracic dissection is a tear in the wall of the aorta, that causes blood to flow between the layers of the aorta and force the layers apart (dissect). This condition is a medical emergency and can quickly lead to death. Since stent grafting has been an effective way to treat other aortic conditions such as aneurysms (bulge in aorta wall), it is believed that the device would be effective in treating dissections. Information will be collected on the performance of the device for 5 years.

ELIGIBILITY:
Inclusion Criteria

* Subject signed an informed consent.
* Subject is at least 18 years old.
* Subject has an acute, complicated Type B aortic dissection with evidence of at least one of the following:
* Malperfusion (visceral, renal, spinal cord and/or lower limb ischemia)
* Visceral ischemia measured by either radiographic or clinical evidence.
* Renal ischemia measured by either radiographic or clinical evidence.
* Spinal cord ischemia measured by either radiographic or clinical evidence.
* Lower limb ischemia measured by either radiographic or clinical evidence.
* Rupture - Measured by radiographic or clinical evidence.
* Subject is hemodynamically stable.
* Subject's anatomy must meet all of the following anatomical criteria:

Proximal landing zone aortic diameter must be between 20 mm and 44 mm;

* Centerline distance from distal margin of left CCA or in cases of bovine anatomy, innominate artery, to start of most proximal tear must be ≥ 20 mm;
* Subject has patent iliac or femoral arteries or can tolerate an iliac conduit that allows endovascular access to the dissection site with the delivery system of the appropriate sized device.
* Thoracic aortic dissection is confirmed, at a minimum, by diagnostic contrast-enhanced computerized tomography angiogram (CTA) with 3-D reconstruction, and/or contrast enhanced magnetic resonance angiogram (MRA) obtained prior to the implant procedure.

Exclusion Criteria

* Planned placement of the COVERED portion of the stent graft over the left carotid artery, or the celiac trunk.
* Subject has systemic infection.
* Subject is pregnant.
* Subject has received a previous stent or stent graft or previous surgical repair in the DTA.
* Subject has had a cerebral vascular accident (CVA) within 2 months.
* Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
* Subject has a history of Marfan Syndrome or other connective tissue disorder.
* Subject is currently participating in an investigational drug or device clinical trial which would interfere with the endpoints and follow-ups of this study.
* Subject has a known allergy or intolerance to the device components.
* Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.
* Subject has a co-morbidity causing expected survival to be less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E. Bavaria, M.D., Principal Investigator — Univ. of Pennsylvania Health System; W. Anthony Lee, M.D., F.A.C.S, Principal Investigator — Lynn Heart Institute, Boca Raton Community Hospital
Locations (17):
- United States (17):
  - USC Keck School of Medicine, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Harbor UCLA, Torrance, California
  - Washington Hospital D.C., Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Northwestern Memorial, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - New York Presbyterian Weill Cornell, New York, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Heart Hospital Medical Center, Dallas, Texas
  - Baylor, Houston, Texas
  - Memorial Hermann Heart and Vascular Institute, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Virginia Commonwealth University MCV Richmond, Richmond, Virginia

REFERENCES:
- [Derived] Bavaria JE, Brinkman WT, Hughes GC, Shah AS, Charlton-Ouw KM, Azizzadeh A, White RA. Five-year outcomes of endovascular repair of complicated acute type B aortic dissections. J Thorac Cardiovasc Surg. 2022 Feb;163(2):539-548.e2. doi: 10.1016/j.jtcvs.2020.03.162. Epub 2020 May 13. PMID 32654872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Started | 50
Completed | 40
Not Completed | 10
Not completed — Death | 8
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 37
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality.
Time Frame: Up to 30 days after the stent graft implant.
Population: Based on number of ITT subjects with available data
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
participants | 4

2. Secondary Outcome: All-cause Mortality
Time Frame: at 12 months
Population: Based on number of ITT subjects with available data. Subjects were considered unevaluable if they were withdrawn before the lower limit of the 12 months follow-up window or were lost to follow-up before the lower limit of the 12 months follow-up window. (One patient withdrew and one was lost to follow-up)
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 48
participants | 7

3. Secondary Outcome: Subjects With Successful Delivery and Deployment of the Device.
Time Frame: At implant.
Population: Based on number of ITT subjects with available data
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
participants | 50

4. Secondary Outcome: Subjects With Coverage of Primary Tear
Time Frame: At implant
Population: Based on number of ITT subjects with available data
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
participants | 50

5. Secondary Outcome: Aortic Rupture
Time Frame: Within 30 days
Population: Based on number of ITT subjects with available data.
Measure: Number; unit: participants
Groups:
- Valiant Thoracic Stent Graft With the Captivia Delivery System: Valiant Thoracic Stent Graft will the Captivia Delivery System: All subjects will be implanted with this device
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
participants | 0

6. Secondary Outcome: Aortic Rupture
Time Frame: Within 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 48
participants | 0

7. Secondary Outcome: Subjects With Secondary Endovascular Procedures
Time Frame: Through12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 48
participants | 4

8. Secondary Outcome: Aortic Remodeling: Subjects With Partial/Complete False Lumen Thrombosis Over the Stented Segment
Time Frame: At 6 months
Population: Based on number of ITT subjects with evaluable imaging data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 33
participants | 25

9. Secondary Outcome: Aortic Remodeling: Subjects With Complete/Partial Thrombosis of the False Lumen Over the Stented Segment
Time Frame: At 12 months
Population: Based on number of ITT subjects with evaluable imaging data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 34
participants | 27

10. Secondary Outcome: Aortic Remodeling: Subjects With Stable (+/- 5mm) or Increase in True Lumen (>5mm) Compared to First Post-procedural CT Over the Stent Graft
Time Frame: at 6 months
Population: Based on number of ITT subjects with evaluable imaging data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 33
participants | 31

11. Secondary Outcome: Aortic Remodeling: Subjects With Stable (+/- 5mm) or Increase in True Lumen (>5mm) Compared to First Post-procedural CT Over the Stent Graft
Time Frame: at 12 months
Population: Based on number of ITT subjects with evaluable imaging data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 34
participants | 32

12. Secondary Outcome: Aortic Remodeling: Subjects With Stable (+/- 5mm) or Decrease in False Lumen (>5mm) Compared to First Post-procedural CT Over the Stent Graft
Time Frame: at 6 months
Population: Based on number of ITT subjects with evaluable imaging data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 33
participants | 25

13. Secondary Outcome: Aortic Remodeling: Subjects With Stable (+/- 5mm) or Decrease in False Lumen (>5mm) Compared to First Post-procedural CT Over the Stent Graft
Time Frame: at 12 months
Population: Based on number of ITT subjects with evaluable imaging data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 34
participants | 28

14. Secondary Outcome: Subjects With Device, Procedure and/or Aortic Related Serious Adverse Events.
Time Frame: at 30 days
Population: Based on number of ITT subjects with available data.
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
participants | 19

15. Secondary Outcome: Subjects With Device, Procedure and/or Aortic Related Serious Adverse Events.
Time Frame: at 12 months
Population: Based on number of ITT subjects with available data. Subjects were considered unevaluable if they were withdrawn or were lost to follow-up before the lower limit of the 12 mos follow-up window.One subject was lost to follow-up and one withdrew before 12 mos. One of these subjects experienced an AE before study exit and was included in the analysis,
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 49
participants | 23

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. Dissection: Medtronic Dissection
Arm/Group | 1. Dissection
Serious Adverse Events (participants affected / at risk) | 23/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Dissection (N=50)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1)
Continued Perfusion from a Branch Vessel requiring Treatment (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1)
Nerve Injury (Injury, poisoning and procedural complications) | 1 (1)
Stent-Graft Endoleak (Injury, poisoning and procedural complications) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 1 (1)
White Blood Cell Count Increased (Investigations) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 3 (3)
Monoplegia (Nervous system disorders) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1)
Spinal Cord Ischaemia (Nervous system disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 2 (2)
Aortic Dissection (Vascular disorders) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1)
Subclavian Artery Embolism (Vascular disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) and institution agree not to publish the results of the study until after the earliest of the following: a)conclusion of the study, b)the early termination of the study, c)at discretion and approval of the sponsor, or d)after sponsor confirms there will be no multicenter study publication, whichever occurs first. PI and institution further agree to submit to sponsor copies of any proposed publication or public presentation at least sixty days before dissemination.